CLINICAL TRIAL: NCT02339935
Title: Improving Hospitalizations for Children With ASD: Testing the Cost and Clinical Efficacy of Integrated Behavioral Intervention
Brief Title: Improving Hospitalizations for Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Kevin Sanders, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 141265
Record Dates: First submitted 2014-12-30; First posted 2015-01-16 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2015-09

CONDITIONS: Autism Spectrum Disorder; Autistic Disorder
Keywords: Autism Spectrum Disorder; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABA Treatment Group (Experimental): 20 Children - 10 hospitalized at Vanderbilt Children's Hospital and 10 hospitalized at Vanderbilt Psychiatric hospital - will receive Brief Analogue Functional Analysis (Brief AFA) targeted to their most problematic behavior(s) while hospitalized
  Interventions: Behavioral: Brief Analogue Functional Analysis
- Control Group (Other): 20 Children - 10 hospitalized at Vanderbilt Children's Hospital and 10 hospitalized at Vanderbilt Psychiatric hospital - will receive all typical standard of care procedures while hospitalized, but will not receive Brief AFA
  Interventions: Other: No Brief AFA

INTERVENTIONS:
Behavioral: Brief Analogue Functional Analysis — The Brief AFA seeks to identify the function of the challenging behavior by creating controlled test conditions in which specific responses are provided for challenging behavior (e.g., attention, escape from task demands, access to tangible - including variants of each as needed), as well as a control condition in which continual access to attention and preferred items is provided. It consists of a 30-90-minute abbreviated analysis comprised of a single exposure to 2-5-minute test and control conditions, along with replication of applicable test conditions and a treatment probe, which provides evidence of challenging behavior function faster than other methods.
  Arms: ABA Treatment Group
Other: No Brief AFA — These participants will receive typical standard of care procedures while hospitalized, but will not receive the additional behavioral intervention
  Arms: Control Group

SUMMARY:
This study aims to implement and test a specific brief Applied Behavior Analysis model for assessing and responding to severe challenging behavior during acute medical and behavioral hospitalization for children with ASD. The investigators will evaluate the impact of this program by conducting a randomized trial across both medical and psychiatric hospital settings.

ELIGIBILITY:
Inclusion Criteria:

* documented diagnosis of an ASD based on clinical DSM-5 diagnostic criteria assessed by attending psychiatrist
* the presence of a significant challenging behaviors (e.g., aggression, property destruction, self-injury, elopement)
* admission to the VPH or medical floors
* individual and caregiver agreement to participate and ability to provide informed consent (and assent).

Exclusion Criteria:

* None

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist | Change from Baseline ABC at Hospital Discharge (an expected average of 42 days) and 3-Months Post-Discharge
  The ABC is a well-validated measure designed to assess for the presence of clinically significant challenging behavior in the areas of irritability and agitation, lethargy and social withdrawal, stereotypic behavior, hyperactivity and noncompliance, and inappropriate speech.
Decrease in Length of Hospitalization | Participants will be followed from admission to discharge, an expected average of 42 days
  Reduction in the days hospitalized past medical clearance).

SECONDARY OUTCOMES:
Clinical Global Impression Scales of Severity | Baseline and Day of Patient's Discharge (an expected average of 42 days from admission)
  Attending physician's impressions of participant's clinical impairment and improvement.
Blinded Observational Ratings | Participants will be followed for duration of hospital stay, an expected average of 42 days
  Blinded coding of the challenging behaviors targeted in the treatment arm
Physician/Nurse/Family Perception of Care | Day of Patient's Discharge (an expected average of 42 days from admission)
  The primary medical attending, lead discharge nurse staff member, and the child's primary parent will also be asked at discharge to provide both quantitative and qualitative ratings of challenges and successes during hospitalization. Caregivers will be contacted to complete a simple interview/questionnaire 3- months post-hospitalization regarding changes in the patient's medication, medical conditions, residential/classroom placement, emergency room visits or psychiatric hospitalizations since the discharge date, as well as ratings of successes implementing components of the behavioral strategies plan utilized during the hospitalization (if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Sanders, MD, Principal Investigator — MEND Clinic - Director
Locations (1):
- Vanderbilt University Medical Center - MEND Clinic, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Sanders K, Staubitz J, Juarez AP, Marler S, Browning W, McDonnell E, Altstein L, Macklin EA, Warren Z. Addressing Challenging Behavior During Hospitalizations for Children with Autism: A Pilot Applied Behavior Analysis Randomized Controlled Trial. Autism Res. 2020 Jul;13(7):1072-1078. doi: 10.1002/aur.2308. Epub 2020 Apr 23. PMID 32329237